CLINICAL TRIAL: NCT03806244
Title: Prospective Study of the Feasibility of Stereotactic Navigation in Laparoscopic Surgery for Colorectal Cancer
Brief Title: Feasibility of Stereotactic Navigation in Laparoscopic Surgery for Colorectal Cancer
Acronym: PELVINAV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the two main investigators
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-002
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: stereotactic navigation; colorectal cancer; laparoscopy; transanal surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREOP (No Intervention): Navigation without intraoperative acquisition of images: Use of conventional preoperative images (CT-MRI) to establish intraoperative navigation.
- PEROP (Experimental): Navigation with intraoperative acquisition of images: Intraoperative acquisition (robotic c-Arm) of images to establish intraoperative navigation.
  Interventions: Other: Intraoperative acquisition (robotic c-Arm) of images

INTERVENTIONS:
Other: Intraoperative acquisition (robotic c-Arm) of images — Conventional laparoscopic colorectal oncologic resection is performed. During the procedure, the operator will identify previously defined anatomical landmarks, point them with an instrument tracked by the navigation system and the accuracy of the stereotactic navigation system will be calculated by comparing the "surgical" anatomical point and its correspondent on the images of the navigation platform.
  Arms: PEROP

SUMMARY:
To evaluate the feasibility and precision of stereotaxic navigation in laparoscopic surgery for colorectal cancer.

DETAILED DESCRIPTION:
* In minimally invasive surgery, the proper identification of the correct anatomical planes can be difficult due to a lack of tactile feedback and the inability to manually palpate the organ prior to resection. Although this can be minimized by careful preoperative planning, the information that can be obtained by images is also of limited utility. Conventional imaging, such as magnetic resonance imaging (MRI) and computed tomography (CT-scan), can provide a detailed view of 2D or 3D internal anatomical structures. However, during surgery, surgeons still have to use their subjective interpretation to translate this information into three-dimensional spatial relationships (ie the patient's actual volume). For this reason, in order to perform adequate resection and avoid injury, the surgeon must constantly infer what is the actual location of the anatomical structures and what is the position of the surgical instruments in relation thereto.
* The proposed study aims to evaluate the feasibility of surgical navigation in patients with colorectal cancer (sigmoid rectum-right-left rectum) and measure its performance in the perspective of a more specific application to rectal cancer approached laparoscopically through the abdomen and / or the anus. The study is proposed to patients with cancer because the measurement of accuracy will be done on predefined anatomical points that will be detectable in the surgical field after oncologic dissection. Benign pathologies do not require this type of extensive dissection and the application of navigation would imply additional risks for patients.
* Surgical navigation will be performed on the basis of preoperative images or intraoperative images.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years old
2. Patient presents with cancer
3. Patient has no contraindication to anesthesia and surgical resection
4. Patient able to receive and understand information about the study and give written informed consent
5. Patient (s) affiliated to the national social security system.

Exclusion Criteria:

1. Patient operated on urgently.
2. Pregnant or lactating patient
3. Patient in an exclusion period (determined by previous or current study).
4. Patient under the protection of justice.
5. Patient under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of Surgical stereotactic navigation defined as the distance, in millimetres, between the position of the surgical landmark and the position determined by the navigation system | up to 7 days post procedure
  Measurement of "accuracy" of surgical navigation defined as the distance measured between the position of "surgical" previously defined anatomical landmarks, pointed with a surgical instrument tracked by the navigation system, and corresponding location of the instrument in the navigation image. A distance equal to or less than 4 mm between the two locations will be considered as an optimum accuracy.

SECONDARY OUTCOMES:
Comparison, in millimeters, of the surgical navigation "accuracy" (as defined in the primary outcome) with or without intraoperative images acquisition | up to 7 days post procedure
  Usefulness of intraoperative images acquisition for the registration process of the navigation system by comparing accuracy of surgical navigation (in mm) with or without intraoperative images acquisition
Difference, in millimetres, between the alignment of the geometric position of the markers in the image space and the actual physical space for stereotaxic navigation | up to 7 days post procedure
  Measurement of "registration error" during surgical navigation defined as the difference between the alignment of the geometric position of the markers in the image space and the actual physical space, with or without intraoperative images acquisition. An error of 2 mm during the recording process will be considered as the optimal parameter
Measurement of the overall operating time (in minutes) with and without intraoperative images acquisition | up to 30 days post procedure
  Evaluation of the impact of the introduction of surgical navigation on the operating time. The measurement of the overall operating time (expressed in minutes), associated with surgical navigation
Measurement of the level of radiation exposure to ionizing factors with and without intraoperative images acquisition | up to 30 days post procedure
  Evaluation of the impact of the introduction of surgical navigation on the exposure of the patient to ionizing radiation, measured with Dose Length Product (DLP) and expressed in mGy * cm
Number of intra and/or postoperative complication | up to 30 days post procedure
  Evaluation of the impact of the introduction of surgical navigation on the incidence of intra- and / or postoperative complications associated with surgical navigation

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Principal Investigator — Service Chirurgie Digestive et Endocrinienne, Nouvel Hôpital Civil de Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marley AR, Nan H. Epidemiology of colorectal cancer. Int J Mol Epidemiol Genet. 2016 Sep 30;7(3):105-114. eCollection 2016. PMID 27766137
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Biondi A, Vacante M, Ambrosino I, Cristaldi E, Pietrapertosa G, Basile F. Role of surgery for colorectal cancer in the elderly. World J Gastrointest Surg. 2016 Sep 27;8(9):606-613. doi: 10.4240/wjgs.v8.i9.606. PMID 27721923
- [Background] Simmonds PC, Primrose JN, Colquitt JL, Garden OJ, Poston GJ, Rees M. Surgical resection of hepatic metastases from colorectal cancer: a systematic review of published studies. Br J Cancer. 2006 Apr 10;94(7):982-99. doi: 10.1038/sj.bjc.6603033. PMID 16538219
- [Background] Rullier E, Sebag-Montefiore D. Sphincter saving is the primary objective for local treatment of cancer of the lower rectum. Lancet Oncol. 2006 Sep;7(9):775-7. doi: 10.1016/S1470-2045(06)70863-4. No abstract available. PMID 16945773
- [Background] Orsini RG, Wiggers T, DeRuiter MC, Quirke P, Beets-Tan RG, van de Velde CJ, Rutten HJ. The modern anatomical surgical approach to localised rectal cancer. EJC Suppl. 2013 Sep;11(2):60-71. doi: 10.1016/j.ejcsup.2013.07.033. No abstract available. PMID 26217114
- [Background] Abu Gazala M, Wexner SD. Re-appraisal and consideration of minimally invasive surgery in colorectal cancer. Gastroenterol Rep (Oxf). 2017 Feb;5(1):1-10. doi: 10.1093/gastro/gox001. Epub 2017 Feb 6. PMID 28567286
- [Background] Bucholz RD. Introduction to Journal of Image Guided Surgery. J Image Guid Surg. 1995;1(1):1-3. doi: 10.1002/(SICI)1522-712X(1995)1:13.0.CO;2-E. No abstract available. PMID 9079420
- [Background] Azagury DE, Dua MM, Barrese JC, Henderson JM, Buchs NC, Ris F, Cloyd JM, Martinie JB, Razzaque S, Nicolau S, Soler L, Marescaux J, Visser BC. Image-guided surgery. Curr Probl Surg. 2015 Dec;52(12):476-520. doi: 10.1067/j.cpsurg.2015.10.001. Epub 2015 Oct 22. No abstract available. PMID 26683419
- [Background] Mezger U, Jendrewski C, Bartels M. Navigation in surgery. Langenbecks Arch Surg. 2013 Apr;398(4):501-14. doi: 10.1007/s00423-013-1059-4. Epub 2013 Feb 22. PMID 23430289
- [Background] Pruliere-Escabasse V, Coste A. Image-guided sinus surgery. Eur Ann Otorhinolaryngol Head Neck Dis. 2010 Mar;127(1):33-9. doi: 10.1016/j.anorl.2010.02.009. Epub 2010 Mar 24. PMID 20822755
- [Background] Risholm P, Golby AJ, Wells W 3rd. Multimodal image registration for preoperative planning and image-guided neurosurgical procedures. Neurosurg Clin N Am. 2011 Apr;22(2):197-206, viii. doi: 10.1016/j.nec.2010.12.001. PMID 21435571
- [Background] Fitzpatrick JM. The role of registration in accurate surgical guidance. Proc Inst Mech Eng H. 2010;224(5):607-22. doi: 10.1243/09544119JEIM589. PMID 20718266
- [Background] Wittmann W, Wenger T, Zaminer B, Lueth TC. Automatic correction of registration errors in surgical navigation systems. IEEE Trans Biomed Eng. 2011 Oct;58(10):2922-30. doi: 10.1109/TBME.2011.2163156. Epub 2011 Jul 29. PMID 21803677
- [Background] Gundle KR, White JK, Conrad EU, Ching RP. Accuracy and Precision of a Surgical Navigation System: Effect of Camera and Patient Tracker Position and Number of Active Markers. Open Orthop J. 2017 May 31;11:493-501. doi: 10.2174/1874325001711010493. eCollection 2017. PMID 28694888
- [Background] Baumhauer M, Feuerstein M, Meinzer HP, Rassweiler J. Navigation in endoscopic soft tissue surgery: perspectives and limitations. J Endourol. 2008 Apr;22(4):751-66. doi: 10.1089/end.2007.9827. PMID 18366319
- [Background] Wijsmuller AR, Romagnolo LGC, Agnus V, Giraudeau C, Melani AGF, Dallemagne B, Marescaux J. Advances in stereotactic navigation for pelvic surgery. Surg Endosc. 2018 Jun;32(6):2713-2720. doi: 10.1007/s00464-017-5968-0. Epub 2017 Dec 6. PMID 29214516
- [Background] Atallah S, Nassif G, Larach S. Stereotactic navigation for TAMIS-TME: opening the gateway to frameless, image-guided abdominal and pelvic surgery. Surg Endosc. 2015 Jan;29(1):207-11. doi: 10.1007/s00464-014-3655-y. Epub 2014 Jun 28. PMID 24972925
- [Background] Atallah S, Martin-Perez B, Larach S. Image-guided real-time navigation for transanal total mesorectal excision: a pilot study. Tech Coloproctol. 2015 Nov;19(11):679-84. doi: 10.1007/s10151-015-1329-y. Epub 2015 Jul 9. PMID 26153411
- [Background] Atallah S, Larach SW, Monson JR. Stereotactic navigation for TAMIS-TME. Minim Invasive Ther Allied Technol. 2016 Oct;25(5):271-7. doi: 10.1080/13645706.2016.1201119. Epub 2016 Jun 27. PMID 27348417
- [Background] Bai M, Liu B, Mu H, Liu X, Jiang Y. The comparison of radiation dose between C-arm flat-detector CT (DynaCT) and multi-slice CT (MSCT): a phantom study. Eur J Radiol. 2012 Nov;81(11):3577-80. doi: 10.1016/j.ejrad.2011.09.006. Epub 2011 Oct 2. PMID 21963617
- [Background] Raman SP, Chen Y, Fishman EK. Evolution of imaging in rectal cancer: multimodality imaging with MDCT, MRI, and PET. J Gastrointest Oncol. 2015 Apr;6(2):172-84. doi: 10.3978/j.issn.2078-6891.2014.108. PMID 25830037
- See also: Image-guided navigation surgery for pelvic malignancies using electromagnetic tracking - Proceedings of the SPIE — http://adsabs.harvard.edu/abs/2016SPIE.9786E..2LN
- See also: Surgical Navigation Systems: A Technological Overview - Conference Paper · June 2014 — https://www.researchgate.net/publication/272787446_Surgical_Navigation_Systems_A_Technological_Overview